CLINICAL TRIAL: NCT02526901
Title: The Born in Guangzhou Cohort Study (BIGCS)
Acronym: BIGCS
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Xiu Qiu, Director of the Born in Guangzhou Cohort Study, Guangzhou Women and Children's Medical Center
Other Study IDs: 2011Y2-00025; 201041-E00741 (Other Grant/Funding Number: Guangzhou Science and Technology Bureau, Guangzhou, China); 2012J5100038 (Other Grant/Funding Number: Guangzhou Science and Technology Bureau, Guangzhou, China); 201508030037 (Other Grant/Funding Number: Guangzhou Science and Technology Bureau, Guangzhou, China)
Record Dates: First submitted 2015-08-13; First posted 2015-08-18 (Estimated); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Intrauterine Hyperglycemia; Pregnancy Outcomes; Neurodevelopment; Immune Development; Childhood Obesity; Host and Microbiome
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During pregnancy: maternal blood, urine and stool. At delivery: cord, cord blood and placenta. During infancy: dry blood spot, stool and blood. Druing childhood: blood, buccal swab and stool.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No treatment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The Born in Guangzhou Cohort Study (BIGCS) was established to investigate the short- and long-term effects of exposure in early life on health consequences in Guangzhou, China. Data are collected regarding environmental, occupational and lifestyle exposures as well as health outcomes in later life. Biological samples including blood and tissue samples are also collected from the participants.

DETAILED DESCRIPTION:
Over the past three decades, China is undergoing rapidly economic development. At the same time, the Western diet and urban lifestyle has been more common than before, which may lead to an increase of incidence of non-communicable chronic diseases, such as diabetes and malignancies. Notably, the current generation of Chinese adults, particularly those in their middle age or older, were born in an era where hardship and rationing was the norm and witnessed a social and epidemiological transition that might have a profound effect on their present health. In contrast, the younger generation is raised in relative material abundance, under the influence of traditional Chinese values such as a strong family orientation and an emphasis on academic success. A birth cohort with would provide an opportunity to examine the short- and long-term effects of exposure in early life on health consequences in this younger generation, in the context of rapid development in China.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with <20 weeks of gestation
* Pregnant women intended to eventually deliver in Guangzhou Women and Children's Medical Center
* Permanent residents or families intended to remain in Guangzhou with their child for ≥3 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women attending their first routine antenatal examinations (usually around week 16) and their partners and offsrping
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-02-01; Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participant with pregnancy outcomes | At delivery
  Including abortion, stillbirth, live birth, preterm birth, low birth weight and birth defects

SECONDARY OUTCOMES:
Neurodevelopment during early childhood | At age of 3 years
  Including adaptive, gross motor, fine motor, language, and social function; assessed using Gesell Developmental Schedules and Ages and Stages Questionnaire
Weight changes during early childhood | At birth, age of 6 weeks, 6 months, 1 year and 3 years
  Weight changes from birth, 6 weeks, 6 months, 1 year to 3 years
Height changes during early childhood | At birth, age of 6 weeks, 6 months, 1 year and 3 years
  Height changes from birth, 6 weeks, 6 months, 1 year to 3 years
Changes of body composition during early childhood | At birth, age of 6 weeks, 6 months, 1 year and 3 years
  Changes of body composition from birth, 6 weeks, 6 months, 1 year to 3 years. Body composition is assessed using Dual Energy X-Ray Absorptiometry

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Qiu, PhD, Principal Investigator — Guangzhou Women and Children's Medical Center, China
Locations (1):
- Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] He JR, Yuan MY, Chen NN, Lu JH, Hu CY, Mai WB, Zhang RF, Pan YH, Qiu L, Wu YF, Xiao WQ, Liu Y, Xia HM, Qiu X. Maternal dietary patterns and gestational diabetes mellitus: a large prospective cohort study in China. Br J Nutr. 2015 Apr 28;113(8):1292-300. doi: 10.1017/S0007114515000707. Epub 2015 Mar 30. PMID 25821944
- See also: BIGCS website — http://113.108.182.54/